CLINICAL TRIAL: NCT04655807
Title: A Phase 2a Randomized, Double-blind, Placebo-controlled, Parallel-group, Multicenter, Proof-of-Concept Clinical Study to Evaluate the Safety and Efficacy of JNJ-64304500 as Add-on Therapy to Standard of Care Biologic Therapy With Anti-Tumor Necrosis Factor Alpha or Anti-Interleukin 12/23 in Responder Not Remitter Participants With Active Crohn's Disease
Brief Title: A Study of JNJ-64304500 as Add-on Therapy in Participants With Active Crohn's Disease
Acronym: DUET
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor Decision.
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR108898; 2020-002701-26 (EudraCT Number); 64304500CRD2002 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2020-11-30; First posted 2020-12-07 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Crohn Disease
MeSH Terms: conditions — Crohn Disease | interventions — Adalimumab; Ustekinumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group 1- Standard of Care (SOC) Biological Therapy: Adalimumab (Experimental): Participants will receive JNJ-64304500 Dose 1 or matching placebo subcutaneous (SC) injection as induction dose (Week 0) followed by JNJ-64304500 Dose 2 or matching placebo SC injection from Week 2 through Week 10 as maintenance dose in addition to adalimumab or its biosimilar as SOC therapy.
  Interventions: Drug: JNJ-64304500; Drug: Placebo; Drug: Adalimumab
- Group 2: SOC Biological Therapy: Ustekinumab (Experimental): Participants will receive JNJ-64304500 Dose 1 or matching placebo SC injection as induction dose (Week 0) followed by JNJ-64304500 Dose 2 or matching placebo SC injection from Week 2 through Week 10 as maintenance dose in addition to ustekinumab as SOC therapy.
  Interventions: Drug: JNJ-64304500; Drug: Placebo; Drug: Ustekinumab

INTERVENTIONS:
Drug: JNJ-64304500 — JNJ-64304500 will be administered as SC injection.
Drug: Placebo — Matching placebo will be administered as SC injection.
Drug: Adalimumab — Adalimumab will be administered as SOC biological therapy.
  Arms: Group 1- Standard of Care (SOC) Biological Therapy: Adalimumab
Drug: Ustekinumab — Ustekinumab will be administered as SOC biological therapy.
  Arms: Group 2: SOC Biological Therapy: Ustekinumab

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of JNJ-64304500 as add-on therapy to standard of care (SOC) biologic treatment with anti-tumor necrosis factor alpha or anti-interleukin 12/23 inhibitors in participants with active Crohn's disease in response but not remission to SOC biologic therapy.

DETAILED DESCRIPTION:
Biologic agents such as anti-tumor necrosis factor (TNF) and interleukin (IL)-12/23 antagonists have become the standard of care (SOC) in the treatment of patients with Crohn's disease. However, many patients fail to fully respond to treatment. This study will evaluate the efficacy of 10 week add on treatment with JNJ-64304500, compared to placebo, in patients taking SOC anti-TNF or anti-IL12/23 biologics. The study consists of a screening phase (up to 8 weeks); treatment phase (up to 12 weeks and follow-up phase (up to 16 weeks after the last administration of study agent). The total study duration will be up to 34 weeks. Key safety assessments include adverse events, clinical laboratory tests (hematology and chemistry), vital signs, monitoring for injection-site and hypersensitivity reactions, and early detection of active tuberculosis.

ELIGIBILITY:
Inclusion Criteria:

* Have confirmed clinical diagnosis of Crohn's disease or fistulizing Crohn's disease of at least 3 months' duration
* Initiated standard of care (SOC) biologic therapy for at least 12 uninterrupted weeks (including the induction dose) prior to Week 0 and agree to continue to maintain their SOC biologic with no change in dose level or interruption for the duration of the study. Adalimumab (including HUMIRA or an equivalent biosimilar which could include: HULIO, HYRIMOZ, IMRALDI, or AMGEVITA) at maintenance dose of 40 milligram (mg) subcutaneous (SC) every 2 weeks (q2w) plus minus (+ -) 4 days or Ustekinumab at maintenance dose of 90 mg SC every 8 weeks (q8w) + - 7 days
* Have active Crohn's disease (CD), with a baseline crohn's disease activity index (CDAI) score of greater than or equal to (>=) 180 but less than or equal to (<=) 400
* Participant with a family history of colorectal cancer, personal history of increased colorectal cancer risk, age greater than (>) 50 years, or other known risk factor must be up-to-date on colorectal cancer surveillance
* Participant who has had extensive colitis for >=8 years, or disease limited to the left side of the colon for >=12 years, must either have had a colonoscopy to assess for the presence of dysplasia within 1 year before the first administration of study agent or a colonoscopy to assess for the presence of malignancy at the screening visit, with no evidence of malignancy
* A woman of childbearing potential must have a negative highly sensitive serum (beta- human chorionic gonadotropin [beta-hCG]) pregnancy test result at screening and a negative urine pregnancy test result at Week 0 and throughout the study

Exclusion Criteria:

* Has complications of Crohn's disease as defined in study protocol
* Currently has or is suspected to have an abscess
* Concomitant or previous medical therapies received: has previously demonstrated suboptimal response, loss of response, or intolerance to more than 2 approved advanced therapies
* Concomitant or previous medical therapies received: corticosteroids and 5-aminosalicylic acid (5-ASA) compounds at unstable or above recommended doses are not permitted. Individuals receiving stable doses (oral corticosteroids at a prednisone-equivalent dose at or below 20 mg/day, or 6 mg/day of budesonide, 2.5 mg/day beclomethasone dipropionate, or at or below 5-ASA doses of 1.5 gram (g)/day) or if individuals have been discontinued, for at least 2 weeks before start of first study intervention (Week 0), are permitted
* Concomitant or previous medical therapies received: has received any of the following prescribed medications or therapies within the specified period or has plans to initiate throughout the study: conventional immunomodulators (that is , azathioprine [AZA], 6-mercaptopurine [6 MP], or methotrexate [MTX]) within 4 weeks of first dose of study intervention; oral immunomodulatory agents (example, 6-thioguanine [6-TG], cyclosporine, tacrolimus, sirolimus, or mycophenolate mofetil, tofacitinib and other Janus kinase [JAK] inhibitors [including investigational JAK inhibitors]) less than (<) 6 weeks or within 5 half-lives of agent before first dose of SOC biologic, whichever is longer; all other immunomodulatory biologic agents (including investigational biologics) received within 12 weeks or within 5 half-lives of first dose of SOC biologic, whichever is longer
* Infections or predisposition to infections criteria: has a stool culture or other examination positive for an enteric pathogen, including clostridium difficile toxin, in the last 4 months unless a repeat examination is negative and there are no signs of ongoing infection with that pathogen
* Has a transplanted organ (with exception of a corneal transplant that needs to have occurred > 12 weeks before screening)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-03-03 (Estimated); Primary Completion 2023-05-24 (Estimated); Study Completion 2023-09-04 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events (AEs) and Treatment Emergent Adverse Events (TEAEs) | Up to Week 26
  An AE can be any unfavorable and unintended sign (including an abnormal finding), symptom, or disease temporally associated with the use of a medicinal (investigational or non investigational) product, whether or not related to that medicinal (investigational or non investigational) product. TEAEs are AEs with onset during the intervention phase or that are a consequence of a preexisting condition that has worsened since baseline.
Number of Participants with Treatment-emergent Serious Adverse Events (SAEs) | Up to Week 26
  TEAEs are AEs with onset during the intervention phase or that are a consequence of a preexisting condition that has worsened since baseline. A SAE is any untoward medical occurrence that at any dose: results in death; is life-threatening; requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent or significant disability/incapacity; is a congenital anomaly/birth defect; is a suspected transmission of any infectious agent via a medicinal product; is medically important.
Number of Participants with TEAEs by System Organ Class with a Frequency Threshold of 5 Percent (%) or More | Up to Week 26
  Number of participants with TEAEs by system organ class with a frequency threshold of 5 % or more will be reported.
Number of Participants with Infections, Serious Infections and Infections Requiring Antimicrobial Treatment | Up to Week 26
  Number of participants with infections, serious infections and infections requiring antimicrobial treatment will be reported.
Number of Participants with Clinically Significant Abnormalities in Vital Signs | Up to Week 26
  Number of participants with clinically significant abnormalities in vital signs will be reported.
Number of Participants with Clinically Significant Abnormalities in Laboratory Tests | Up to Week 26
  Number of participants with clinically significant abnormalities in laboratory tests will be reported.
Number of Participants with AEs Leading to Treatment Discontinuation | Up to Week 26
  Number of participants with AEs leading to treatment discontinuation will be reported.
Change from Baseline in the Crohn's Disease Activity Index (CDAI) Score at Week 12 | Baseline and Week 12
  Change from baseline in the CDAI score at Week 12 will be reported. CDAI will be assessed by collecting information on 7 different Crohn's disease-related variables (extra-intestinal manifestations, abdominal mass, weight, hematocrit, total number of liquid or very soft stools, abdominal pain/cramping and general well-being) with scores ranging from 0 to approximately 600. The last 4 variables are scored over 7 days by the participant in a diary. A decrease in CDAI over time indicates improvement in disease activity.

SECONDARY OUTCOMES:
Percentage of Participants Achieving Clinical Response | Week 12
  Percentage of participants achieving a clinical response as measured by CDAI score (including greater than or equal to [>=] 50, >=70, >=100, and >=150 point reduction from baseline in CDAI) will be reported.
Percentage of Participants Achieving Clinical Remission | Week 12
  Percentage of participants achieving a clinical remission as measured by CDAI score (CDAI less than [<] 150) will be reported.
Change from Baseline in the Simple Endoscopic Score for Crohn's disease (SES-CD) at Week 12 | Baseline and Week 12
  Change from baseline in the SES-CD score at Week 12 will be reported. The SES-CD score is based on the evaluation of 4 endoscopic components (presence/size of ulcers, proportion of mucosal surface covered by ulcers, proportion of mucosal surface affected by any other lesions, and presence/type of narrowing/strictures) across 5 ileocolonic segments. Each endoscopic component is scored from 0 to 3 for each segment, and a total score is derived from the sum of all the component scores (range, 0 to 56).
Percentage of Participants Achieving an Endoscopic Response | Week 12
  Percentage of participants achieving an endoscopic response defined as at least a 50% improvement from baseline in the SES-CD.
Percentage of Participants Achieving an Endoscopic Remission | Week 12
  Percentage of participants achieving an endoscopic remission defined as an SES-CD score less than or equal to (<=) 2.
Change From Baseline in Abdominal Pain (AP) | Baseline up to Week 12
  Change in AP from baseline based on a 0 to 10 numerical rating scale (NRS) will be reported. A score of 0 represents "no abdominal pain" and a score of 10 represents the "worst possible AP," with greater scores indicating greater pain severity and intensity.
Percentage of Participants Achieving Patient-Reported Outcome (PRO)-2 Remission | Week 12
  Percentage of participants achieving a PRO-2 remission defined as AP mean daily score (AP component of the CDAI score) at or below 1 and stool frequency (SF) mean daily score at or below 3, that is, AP <=1 and SF <=3.
Serum Concentrations of JNJ-64304500 | Up to Week 26
  Serum concentrations of JNJ-64304500 will be reported.
Number of Participants with Antibodies to JNJ-64304500 | Up to Week 26
  Antibody titers binding to JNJ-64304500 in positive samples will be reported.
Number of Participants with Neutralizing Antibodies to JNJ-64304500 | Up to Week 26
  Number of participants receiving at least one dose of JNJ-64304500 with neutralizing antibodies to JNJ-64304500 will be summarized.
Change in Pharmacodynamics (PD) Biomarker Levels of C-Reactive Protein (CRP) from Baseline Compared with Placebo | Baseline, up to Week 26
  Change in PD biomarker levels of CRP from baseline compared with placebo will be reported.
Change in PD Biomarker Levels of Fecal Calprotectin from Baseline Compared with Placebo | Baseline, up to Week 26
  Change in PD biomarker levels of fecal calprotectin from baseline compared with placebo will be reported.
Change in PD Biomarker Levels of Fecal Lactoferrin from Baseline Compared with Placebo | Baseline, up to Week 26
  Change in PD biomarker levels of fecal lactoferrin from baseline compared with placebo will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Medisphere Medical Research Center, Llc, Evansville, Indiana, United States

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency

REFERENCES:
- [Derived] Hasskamp J, Meinhardt C, Timmer A. Anti-IL-12/23p40 antibodies for induction of remission in Crohn's disease. Cochrane Database Syst Rev. 2025 May 13;5(5):CD007572. doi: 10.1002/14651858.CD007572.pub4. PMID 40357993